CLINICAL TRIAL: NCT03323853
Title: The Utility of the Computerized Assessment and Referral System (CARS) Screener for Mental Health Evaluations in the Emergency Setting
Brief Title: Computerized Assessment and Referral System Screener for Mental Health Evaluations in the Emergency Setting
Acronym: CARS-SA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 206914
Record Dates: First submitted 2017-10-17; First posted 2017-10-27 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Automobiles

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARS-SA Report (Experimental): Emergency care providers for subjects in this group will receive a copy of the subject's CARS-SA summary results.
  Interventions: Behavioral: Computerized Assessment and Referral System (CARS) Self-Assessment Screener; Behavioral: CARS-SA Summary Results
- No CARS-SA Report (Other): Emergency care providers for subjects in this group will not receive a copy of the subject's CARS-SA summary results.
  Interventions: Behavioral: Computerized Assessment and Referral System (CARS) Self-Assessment Screener

INTERVENTIONS:
Behavioral: Computerized Assessment and Referral System (CARS) Self-Assessment Screener — Subjects will take the CARS-SA Screener.
  Other Names: CARS-SA Screener
Behavioral: CARS-SA Summary Results — Subjects will be evaluated by emergency care providers using the CARS-SA Summary Results Report.
  Other Names: CARS-SA Report
  Arms: CARS-SA Report

SUMMARY:
This is a hybrid effectiveness-implementation randomized controlled trial which will be conducted at the emergency department (ED) at the University of Arkansas for Medical Sciences (UAMS) in Little Rock, Arkansas.

The hypothesis of this study is that use of the CARS (a computerized mental health screener) will modify emergency department treatment of patients with previously undiagnosed mental illness.

DETAILED DESCRIPTION:
This pragmatic mixed methods clinical trial will compare the intervention of providing a CARS screener report to emergency providers to not providing the report. It will also collect qualitative data regarding implementation of the CARS screener and report. Consecutive patients presenting when a research associate is available will be approached to participate. Patients will be approached after evaluation by an emergency physician.

The Computerized Assessment and Referral System (CARS) is based on the Composite International Diagnostic Interview (CIDI), a validated instrument for assessing mental health diagnoses.CARS was piloted at 6 different sites in 2016, all in DUI populations. As CARS has not been specifically validated on non-DUI populations, investigators will collect alcohol history (see below). The CARS self-assessment version (CARS-SA) will be utilized in this study.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Not incarcerated
* English-speaking and English-writing (as translators will not be available for this study)

Exclusion Criteria:

* Unable or unwilling to complete CARS screener
* Unable or unwilling to provide any history of alcohol abuse
* Currently presenting with a chief complaint of a psychiatric symptom
* Currently presenting with a substance use complaint
* History of a known psychiatric condition
* Patients taking psychiatric medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2017-12-30 (Actual); Primary Completion 2019-12-21 (Actual); Study Completion 2019-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Wilson, M.D., Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson RG Jr, Mullinax S, De Monte R, McBain S, Porter A, Eastin C, Landes SJ, Wilson MP. Effectiveness of a Self-Administered Computerized Mental Health Screening Tool in the Emergency Department. Psychiatr Serv. 2023 Nov 1;74(11):1180-1184. doi: 10.1176/appi.ps.20220523. Epub 2023 May 10. PMID 37161345

RESULTS

PARTICIPANT FLOW:
Groups:
- CARS Report: CARS Report: Patients will be evaluated by emergency providers using the CARS report
- No CARS Report: No CARS Report: Patients will be evaluated by emergency providers without using the CARS report
Period: Overall Study
Arm/Group | CARS Report | No CARS Report
Started | 213 | 238
Completed | 213 | 238
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CARS Report | No CARS Report | Total
Number analyzed (Participants) | 213 | 238 | 451
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.28 (16.23) | 40.79 (15.45) | 40.55 (15.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 121 | 145 | 266
  Male | 92 | 93 | 185
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With CARS Mental Health Diagnoses Made in the ED; the Number of Psychiatry Evaluations in the Emergency Department (ED); and the Number of Mental Health Referrals Made From the ED
Description: The composite measure includes: the number of CARS mental health diagnoses made in the ED; the number of psychiatry evaluations in the emergency department (ED); and the number of mental health referrals made from the ED.
Time Frame: Up to 12 hours
Measure: Count of Participants; unit: Participants
Arm/Group | CARS Report | No CARS Report
Number analyzed (Participants) | 213 | 238
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Duration of ED visit (typically 2 hours)
Arm/Group | CARS Report | No CARS Report
All-Cause Mortality (participants affected / at risk) | 0/213 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/238
Other Adverse Events (participants affected / at risk) | 0/213 | 0/238

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03323853/Prot_SAP_000.pdf